CLINICAL TRIAL: NCT03841864
Title: A Comparison of Traditional Technique Peripheral Intravenous [PIV] Catheter Insertion to the Utilization of Ultrasound Guidance for the Development of a Vein Classification System and Difficult IV Insertion Algorithm. A Prospective Observational Study
Brief Title: Ultrasound Guided Peripheral IV Insertion
Acronym: USGPIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Anesthesia Program Director, M.D, PhD, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00054941
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: This study will partition all CSMC elective pre-operative patients into grade 1, 2a, 2b and 3 classifications to better assess the patient population distribution. Grade 2A vein classification cohort 2nd IV insertion attempt success rate comparison of traditional vs ultrasound guided technique, IV insertion pain scores and patient satisfaction, will be compared amongst the 2 different modalities for peripheral IV insertion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Grade 1 Vein Visualization (Other): Visual vein classification grade described as excellent Visualization. Objective vein criteria to be included in this group are vein raised above skin and wider than 1mm. Initial IV placement will be traditional attempt but subsequent attempts will be provider discretion for traditional vs ultrasound guided placement
  Interventions: Other: IV placement using ultrasound guidance vs traditional method
- Grade 2A Vein Visualization (Other): Veins that don't fit grade 1 or 2b classification (see respective group descriptions). This groups visual vein classification is described as fair visualization. Initial IV placement will be traditional attempt but subsequent attempts will be provider discretion for traditional vs ultrasound guided placement
  Interventions: Other: IV placement using ultrasound guidance vs traditional method
- Grade 2b Vein Visualization (Other): Only faint vein shadow appearance described as poor visualization. Initial IV placement attempt will be ultrasound guided
  Interventions: Other: IV placement using ultrasound guidance vs traditional method
- Grade 3 Vein Visualization (Other): No vein visualization. Initial IV placement attempt will be ultrasound guided
  Interventions: Other: IV placement using ultrasound guidance vs traditional method

INTERVENTIONS:
Other: IV placement using ultrasound guidance vs traditional method — Ultrasound guided IV placement

SUMMARY:
Hypothesis The initial use of ultrasound guidance when indicated for difficult peripheral IV access will reduce the number of attempts required to achieve successful peripheral IV insertion and improve patient care and satisfaction.

DETAILED DESCRIPTION:
Study objective The purpose of this research study is to compare 2 established peripheral IV insertion techniques (traditional vs ultrasound guided) in order to develop an algorithmic approach to peripheral IV insertion. Patient characteristics, medical history and co-morbidities, in addition to a pre-insertion physical exam vein assessment, will allow for the introduction of a vein classification system and a difficult IV insertion algorithm. Selecting the optimal modality for initial IV insertion will decrease the total number of attempts, facilitate appropriate gauge and location of IV insertion, avoid central line placement, decrease IV insertion pain scores and improve patient satisfaction. Currently, ultrasound guided peripheral IV insertion is performed by the IV team at Cedars-Sinai Medical Center or a trained anesthesia provider as a rescue technique after multiple failed attempts by traditional technique. Secondary to the constraints of both trained providers and equipment resources, the cohort of difficult IV insertion patients are subjected to multiple traditional IV insertion attempts prior to escalation to ultrasound guidance and occasionally, unnecessary central line placements indicated by only poor intravenous access.

Primary end point: Grade 2A vein classification cohort 2nd IV insertion attempt success rate comparison of traditional vs ultrasound guided technique, IV insertion pain scores, Patient satisfaction Secondary end points: Grade 2B and grade 3 vein classification ultrasound guided IV insertion success rate. Grade 1 and 2a vein classification 1st attempt IV insertion success rate. Grade 1 visualization 2nd attempt IV insertion success rate comparison of traditional vs ultrasound guided technique. Difficult IV insertion risk factors and associations, IV gauge and location, central line placement because of inadequate peripheral IV access

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring pre-operative IV

Exclusion Criteria:

* Emergency Surgery, patient refusal, non-english speaking (USGPIV modality available to them but time restrictive to consent for study), pediatrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Grade 1 and Grade 2A vein classification cohort 2nd IV insertion attempt success rate comparison of traditional vs ultrasound guided technique | 9 months after patient recruitment begins
  IV insertion success rate comparison on the second IV insertion attempt (after after 1x unsuccessful IV insertion using traditional technique) between traditional technique versus ultrasound guidance for grade 1 and 2a visual vein classification grades. For an 80% powered study to detect a 30% difference in success rate, an N of 50 is required in each group. Outcome will be successful vs unsuccessful IV insertion

SECONDARY OUTCOMES:
Grade 2B and Grade 3 vein classification IV placement success rate | 9 months after patient recruitment begins
  Ultrasound IV insertion success rate for grade 2B and grade 3 using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, M.D., PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Final vein classification system and difficult IV algorithm. We will publish success rates of different modalities on different vein grades

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736